CLINICAL TRIAL: NCT00541021
Title: Phase III Randomized, Double-blind Study Comparing Gemcitabine and Sorafenib or a Placebo in Patients With Locally Advanced or Metastatic Cancer of the Pancreas.
Brief Title: Gemcitabine With or Without Sorafenib in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000564099; IPC-BAYPAN; INCA-RECF0426; IPC-2005-006
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-07

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; stage IV pancreatic cancer; adenocarcinoma of the pancreas; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Sorafenib

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: sorafenib tosylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether giving gemcitabine together with sorafenib is more effective than giving gemcitabine alone in treating pancreatic cancer.

PURPOSE: This randomized phase III trial is studying giving gemcitabine together with sorafenib to see how well it works compared with giving gemcitabine alone in treating patients with locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare progression-free survival.

Secondary

* Compare toxicities.
* Compare response rate.
* Compare overall survival.
* Evaluate clinical benefits.
* Compare quality of life.
* Identify biomarkers that predict therapeutic response.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral sorafenib tosylate twice daily and gemcitabine hydrochloride IV once weekly for 7 weeks followed by 1 week of rest (course1). For the next 2 courses, patients receive gemcitabine hydrochloride weekly for 3 weeks followed by 1 week of rest and sorafenib tosylate twice daily.
* Arm II: Patients receive oral placebo twice daily and gemcitabine hydrochloride as in arm I.

After completing 3 courses of therapy, patients in both arms who have stable or responding disease may continue to receive sorafenib tosylate or placebo in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Diagnosis of adenocarcinoma of the pancreas

  * Locally advanced or metastatic disease
* Measurable disease, defined as at least 1 lesion measurable by RECIST criteria

Exclusion criteria:

* Brain metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* WHO performance status 0-2
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Creatinine < 1.5 times normal
* Transaminases < 2 times normal (5 times normal if liver metastases)
* Total bilirubin < 1.5 times normal
* Fertile patients must use effective contraception

Exclusion criteria:

* Pregnant or nursing
* Intestinal occlusion
* Prior inflammatory intestinal disease
* Crohn's disease
* Hemorrhagic rectal colitis
* Peripheral neuropathy > grade 2
* Other severe illness, including any of the following:

  * Unstable cardiac disease, even if treated
  * Psychological or neurological disease including dementia
  * Uncontrolled active infection
  * Other severe illness that would compromise study participation
* Impossible to receive study therapy due to geographical, social, or psychological reasons
* Other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics
* At least 6 months since prior chemotherapy or radiochemotherapy
* At least 4 weeks since prior radiotherapy and/or surgery

Exclusion criteria:

* Prior therapy for advanced disease
* Prior inhibitors of kinase signaling (e.g., ras/raf, MEK, AKT, mTOR, or farnesyl transferase)
* Prior inhibitors of angiogenesis (e.g., bevacizumab)
* Prior organ graft or allogeneic transplantation
* Prior extensive intestinal resection
* Concurrent participation in another therapeutic study
* Concurrent inductors of CYP3A4 (e.g., barbiturates, anti-epileptics, or rifampicin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Toxicities
Response rate
Overall survival
Clinical benefits
Quality of life by QLQ-C30
Biomarkers of response

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Viret, MD — Institut Paoli-Calmettes
Locations (1):
- Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille, France